CLINICAL TRIAL: NCT04778228
Title: Driving Pressure as a Predictor of Mortality in Acute Respiratory Distress Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shahenda Mohamed gamal eldin mohamed ali, principle investigator (assistant lecturer at Assiut university), Assiut University
Other Study IDs: driving pressure in ARDS
Record Dates: First submitted 2021-02-13; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: ARDS
Keywords: Driving pressure
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: mechanical ventilation — critically ill patients requiring mechanical ventilation (MV) were ventilated using high tidal volumes (Vt) and high airway pressures, until the pivotal ARDS net randomized controlled trial (RCT) demonstrated that a "lung-protective" MV strategy using a Vt of 4-8 mL/kg predicted body weight (PBW) and moderate levels of positive end-expiratory pressure (PEEP) improved survival (2). Since then, limitation of Vt to 4-8 mL/kg PBW, plateau pressures (Pplat) to a maximum of 30 cm H2O, and application of PEEP 10 -16 cm H2O represent the standard for MV in ARDS patients.
  Other Names: protective lung strategy

SUMMARY:
The aim of this study is to make analysis of potentially modifiable factors contributing to outcome of mechanically ventilated ARDS adult patient receiving lung protective strategy.

Primary Objective: is to evaluate whether DP was superior to the variables that define it in predicting hospital outcome including mortality.

Secondary Objective: is to identify manageable factors associated with outcome such as ventilator-related parameters and to investigate the role of non-modifiable factors such as demographic characteristics, severity of illness.

DETAILED DESCRIPTION:
The acute respiratory distress syndrome (ARDS) is an acute and intense inflammatory disease process of the Lungs, characterized clinically by severe hypoxemia and bilateral pulmonary infiltrates. The hospital mortality ranges between 35% and 45% (1). Traditionally, critically ill patients requiring mechanical ventilation (MV) were ventilated using high tidal volumes (Vt) and high airway pressures, until the pivotal ARDS net randomized controlled trial (RCT) demonstrated that a "lung-protective" MV strategy using a Vt of 4-8 mL/kg predicted body weight (PBW) and moderate levels of positive end-expiratory pressure (PEEP) improved survival (2).

The driving pressure (DP) (calculated as the Pplat minus applied PEEP) has been suggested as a major determinant for the beneficial effects of the three main components of lung-protective MV, namely, Vt, Pplat, and PEEP. and also a given DP would have different effects on outcome depending on the Vt, Pplat, and PEEP (3).

A retrospective analysis of several trials in patients with ARDS comparing different PEEP levels at the same VT or different VT levels at the same PEEP, or a combination of both, found that ΔPrs is the stronger predictor of mortality as compared with Pplats (3).

ELIGIBILITY:
Inclusion Criteria:

* ARDS Patients: who are treated with lung-protective MV and assessed on standardized ventilatory settings(4) at 24 hours after ARDS onset . All patients will meet the American-European Consensus Conference criteria for ARDS (5) on PEEP greater than or equal to 5 cm H2O and Berlin criteria for moderate or severe ARDS (6).

Exclusion Criteria:

* Patients with left atrial hypertension, as diagnosed by the attending physician, as the primary cause of respiratory failure.
* Anticipated duration of mechanical ventilation of less than 48 hours.
* Severe chronic respiratory disease; neuromuscular disease that would prolong mechanical ventilation.
* Intracranial hypertension; morbid obesity; pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  ARDS Patients: who are treated with lung-protective MV and assessed on standardized ventilatory settings(4) at 24 hours after ARDS onset . All patients will meet the American-European Consensus Conference criteria for ARDS (5) on PEEP greater than or equal to 5 cm H2O and Berlin criteria for moderate or severe ARDS (6).
  Exclusion criteria:
  * Patients with left atrial hypertension, as diagnosed by the attending physician, as the primary cause of respiratory failure.
  * Anticipated duration of mechanical ventilation of less than 48 hours.
  * Severe chronic respiratory disease; neuromuscular disease that would prolong mechanical ventilation.
  * Intracranial hypertension; morbid obesity; pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
driving pressure | during intubation UP TO 28 days
  more than or less than 14 cmH2O

SECONDARY OUTCOMES:
ventilator free days and hospital stay. | 28 days
  correlate the driving pressure level with the number of days free of ventilator and earlier hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt